CLINICAL TRIAL: NCT02229045
Title: Phase II Study of Albumin Bound Paclitaxel With 5-FU and CF as Second Line in Taxanes Naive Advanced Gastric Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Ruihua Xu, Professor of Medical Oncology,Vice-president of Sun Yat-sen University Cancer Center, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ABI-FU
Record Dates: First submitted 2014-03-08; First posted 2014-08-29 (Estimated); Last update posted 2014-08-29 (Estimated); Status verified 2014-08

CONDITIONS: Gastric Caner
Keywords: gastric caner; Albumin Bound Paclitaxel; 5-FU/CF; taxanes naive
MeSH Terms: interventions — Albumin-Bound Paclitaxel; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Albumin Bound Paclitaxel With 5-FU/CF (Experimental): Albumin Bound Paclitaxel 150 mg/m2 (on day 1),5FU 400 mg/m2 iv d1, 2.4g/ m2 civ,d1-d3 every 2 weeks until disease progress or intolerable toxicity.
  Interventions: Drug: Albumin Bound Paclitaxel; Drug: 5-FU

INTERVENTIONS:
Drug: Albumin Bound Paclitaxel — Albumin Bound Paclitaxel 150 mg/m2 (on day 1), every 2 weeks until disease progress or intolerable toxicity.
  Other Names: Abraxane
Drug: 5-FU — 5-FU 400 mg/m2 iv d1, 2.4g/ m2 civ,d1-d3 every 2 weeks until disease progress or intolerable toxicity.

SUMMARY:
The purpose of this study is to evaluate the effectiveness and safety of albumin bound paclitaxel plus 5-FU and as second-line therapy in the treatment of taxanes naive patients with advanced gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma of the stomach with inoperable locally advanced or recurrent and/or metastatic disease.
* Male or female.
* Age 18 -75.
* Previous one line of non-taxane chemotherapy for advanced/metastatic disease.
* Measurable disease, according to the Response Evaluation Criteria in Solid Tumours(RECIST)
* ECOG Performance status 0, 1 or 2
* Haematological, Biochemical and Organ Function: Neutrophil count >2.0 × 10 9/L, platelet count > 100 ×10 9/L. Serum bilirubin< 1.5 × upper limit of normal (ULN); or, AST or ALT < 2.5 × ULN (or < 5 × ULN in patients with liver metastases); or, alkaline phosphatase< 2.5 × ULN (or > 5 × ULN in patients with liver metastases,Creatinine clearance > 60 mL/min.
* Signed informed consent.

Exclusion Criteria:

* No prior chemotherapy for gastric cancer.
* Received any investigational drug treatment within 30 days of start of study treatment.
* Patients with active gastrointestinal bleeding.
* Neurological toxicity ≥ grade 2 NCI-CTCAE.
* Other malignancy within the last 5 years, except for carcinoma in situ of the cervix, or basal cell carcinoma.
* History or clinical evidence of brain metastases.
* Serious uncontrolled systemic intercurrent illness, e.g. infections or poorly controlled diabetes.
* Pregnancy women.
* Subjects with reproductive potential not willing to use an effective method of contraception.
* Patients with known active infection with HIV.
* Known hypersensitivity to any of the study drugs

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Estimated)
Dates: Start 2010-11; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
PFS(Progression-free survival ) | 80% PFS events,, an expected average of 10 months
  The PFS was calculated from the initiation of chemotherapy to the date of disease progression or death

SECONDARY OUTCOMES:
OS (Overall survival ) | OS follow-up period: 18 months or 80% OS events, whichever occurs first
  Overall survival was measured from the initiation of chemotherapy to the date of the last follow-up or death.

OTHER OUTCOMES:
ORR (Overall tumor response) | 80% PFS events, an expected average of 10 months
  Overall tumor response: This is defined as the occurrence of either a confirmed complete (CR) or a partial (PR) best overall response as determined by the RECIST criteria from confirmed radiographic evaluations of target and non-target lesions.

CONTACTS AND LOCATIONS:
Overall Officials: Ruihua Xu, PhD,MD, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China